CLINICAL TRIAL: NCT01383850
Title: NCPAP + Heliox as a Treatment for Infant Respiratory Distress Syndrome (RDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Prof. Fabio Mosca, Fondazione Ospedale Maggiore Policlinico Milano
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Heliox
Record Dates: First submitted 2011-03-09; First posted 2011-06-28 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Respiratory Distress Syndrome; Bronchopulmonary Dysplasia
Keywords: preterm infants; nasal continuous positive airway pressure; heliox; bronchopulmonary dysplasia.
MeSH Terms: conditions — Respiratory Distress Syndrome; Bronchopulmonary Dysplasia | interventions — heliox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NCPAP + standard air (Active Comparator)
  Interventions: Other: NCPAP + standard air; Other: NCPAP + Heliox
- NCPAP + Heliox (Experimental)
  Interventions: Other: NCPAP + standard air; Other: NCPAP + Heliox

INTERVENTIONS:
Other: NCPAP + standard air — NCAP (SiPAP, Vyasis) was used to administer standard air
Other: NCPAP + Heliox — Heliox21 (mixture of Helium 80%- Oxygen 20%) (BOC Medical UK- The Linde group) was stored in 10 liter cylinders and administrated through NCPAP for 12 hours (study period) starting from randomization.

SUMMARY:
Infants born between 28 and 32 weeks' gestation with radiological findings and clinical symptoms of moderate RDS, requiring respiratory support with Nasal Continuous Positive Airway Pressure (NCPAP) within the first hour of life, were randomized to receive either standard medical air or a Heliox/Oxygen mixture 80/20 (Heliox) during the first 12 hours of life, followed by medical air until NCPAP was needed. The aim of the study was to assess the therapeutic effects of breathing a low-density gas mixture (heliox: 80% helium and 20% oxygen) in premature babies with Respiratory Distress Syndrome (RDS), undergoing NCPAP in terms of reducing the rate of mechanical ventilation (MV).

ELIGIBILITY:
Inclusion Criteria:

* inborn infants between 28 and 32 weeks of GA
* Silverman score > 5,
* radiological finding of RDS
* a requirement of inspiratory flow of oxygen (FiO2) > 0,25 (SaO2 ) between 88-95% within the first hour of life.

Exclusion Criteria:

* major congenital malformations
* intraventricular hemorrhage (IVH) more than grade 2
* need of intubation in the delivery room or requirement of FiO2 >0,4 during the first hour of life.

Ages: 28 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2008-02; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Efficacy in reducing need of MV | 7 days
  efficacy in reducing need of intubation for MV in infantans undergoing NCPAP within the first 7 days of life

SECONDARY OUTCOMES:
surfactant need | participants will be followed for the duration of hospital stay, an expected average of 10 weeks
  number of doses of exogenous surfactant
major complications of prematurity | participants will be followed for the duration of hospital stay, an expected average of 10 weeks
  incidence of major complications of prematurity
ventilatory assistance | participants will be followed for the duration of hospital stay, an expected average of 10 weeks
  number of days of ventilatory assistance
length of stay | participants will be followed for the duration of hospital stay, an expected average of 10 weeks
  number of days of hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- NICU, Fondazione IRCCS Cà Granda - Ospedale Maggiore Policlinico, Università degli Studi di Milano, Milan, Italy

REFERENCES:
- [Derived] Colnaghi M, Pierro M, Migliori C, Ciralli F, Matassa PG, Vendettuoli V, Mercadante D, Consonni D, Mosca F. Nasal continuous positive airway pressure with heliox in preterm infants with respiratory distress syndrome. Pediatrics. 2012 Feb;129(2):e333-8. doi: 10.1542/peds.2011-0532. Epub 2012 Jan 30. PMID 22291116